CLINICAL TRIAL: NCT06742905
Title: Echocardiographic Acquisition With Geographic Separation of Patients and Sonographers With Roboot Assistance (EAGER)
Brief Title: Echo Acquisition Despite Geographic Separation by Replication of Human Movements (EAGER)
Acronym: EAGER
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baker Heart and Diabetes Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Diagnostic
Other Study IDs: BakerHeartDiabetesI
Record Dates: First submitted 2024-12-16; First posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Echocardiography
Keywords: Echocardiography

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard echo (Active Comparator): Standard echo exam provided by a sonographer using a standard view template
  Interventions: Diagnostic Test: Standard echocardiogram
- Robotic echo (Experimental): Robotic echo exam provided by a sonographer using a standard view template
  Interventions: Diagnostic Test: Robot-guided echo

INTERVENTIONS:
Diagnostic Test: Robot-guided echo — This echo will be performed by a remote sonographer, though a robot
  Arms: Robotic echo
Diagnostic Test: Standard echocardiogram — Echocardiogram acquired by a sonographer at the patient's bedside
  Arms: Standard echo

SUMMARY:
Echocardiography is a cornerstone of modern cardiology management, but access in rural and remote areas is limited. We have developed a robot ("Edler" named after the originator of echocardiography) which enables a sonographer to complete an examination at a distance. This study seeks to compare the images obtained by both methods, the completeness of the exam over a feasible time, and to identify particular components of the exam that are difficult to obtain using the robot.

DETAILED DESCRIPTION:
The EAGER study is an effectiveness and feasibility trial of robot -assisted echo.

Patients who have undergone a standard echo will be asked to have a repeat study with a different sonographer, working remotely, obtaining images using the robot. This study is limited to 1 hour and as many views as possible will be obtained. During the study, the remote sonographer and patient are in direct contact over a video link. Another person will be in the room with the patient and the patient will be instructed on the use of a stop switch which will disengage the robot if they feel uncomfortable.

The acquired images will be saved to the imaging cloud and interpreted by an imaging specialist blinded to the original echocardiogram. A side-by-side comparison will be undertaken for each view, and image quality and study completeness will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Having a conventional echocardiogram

Exclusion Criteria:

* Declined consent to undergo both examinations

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion complete | 1 hour
  Proportion of a standard acquisition protocol obtainable using robotic acquisition over 1 hour

SECONDARY OUTCOMES:
Proportion complete | 1 hour
  Proportion of echo views with the same information provided by conventional echo
Proportion diagnostic features correctly identified by robotic echo | 1 hour
  Proportion diagnostic features correctly identified by robotic echo

CONTACTS AND LOCATIONS:
Locations (1):
- Baker Heart and Diabetes Institute, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data that underlie the results reported in this project (text, tables, figures and appendices) will be made available.
Supporting Information: Study Protocol
Time Frame: Dates - material will be made available immediately following publication, with no end date.
Access Criteria: The authors are pleased to collaborate with other researchers who provide a methodologically sound proposal, to achieve the aims of the approved proposal, including individual participant data meta-analysis.
  Proposals should be directed to tom.marwick@baker.edu.au. To gain access, data requestors will need to sign a data access agreement.
URL: https://www.baker.edu.au/research/laboratories/imaging-research